CLINICAL TRIAL: NCT00228462
Title: A 1-year, Multicenter, Randomized, Double-blind, Parallel Group, Placebo-controlled Phase 3 Study to Evaluate Prevention of Relapse in Patients in Stable Chronic Schizophrenia Receiving Either Sustained-release Quetiapine Fumarate (SEROQUEL) or Placebo (Abbreviated)
Brief Title: Relapse Prevention, RoW: Study to Evaluate Prevention of Relapse in Patients in Stable Chronic Schizophrenia Receiving Either Seroquel or Placebo
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1444C00004
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2013-01-04 (Estimated); Status verified 2013-01

CONDITIONS: Schizophrenia
Keywords: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Drug: Seroquel (quetiapine)

SUMMARY:
This study is being carried out to see if quetiapine (Seroquel) is effective in preventing patients from a schizophrenic relapse when studied for a long time (1 year) and if so, how it compares with non-active treatment.

ELIGIBILITY:
Inclusion Criteria:

* Stable schizophrenic patients who have provided written informed consent
* Patients 18 to 65 years old who remain clinically stable after switching to a stable dose of Seroquel (quetiapine).

Exclusion Criteria:

* Patients with risk of suicide, other disorders or substance abuse that might interfere with the patient's ability to co-operate,
* Expected non-compliance to treatment
* Known diabetes mellitus,
* Contraindications,
* Intolerance or non-responsiveness to Seroquel or other safety issues.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2005-03; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
The primary objective in this study is to demonstrate superior efficacy of quetiapine to placebo by evaluating relapse prevention in long-term use in patients with schizophrenia as measured by the time to first psychiatric relapse up to one year

SECONDARY OUTCOMES:
To demonstrate superiority of quetiapine to placebo by evaluating the risk of relapse in long-term use in patients with schizophrenia by evaluating the one-year relapse rate

CONTACTS AND LOCATIONS:
Overall Officials: AstraZeneca Seroquel Medical Science Director, MD, Study Director — AstraZeneca
Locations (5):
- Bulgaria (3):
  - Investigative Site, Burgas
  - Investigative Site, Radnevo
  - Investigative Site, Sofia
- Poland (2):
  - Investigative Site, Bydgoszcz
  - Investigative Site, Tuszyn